CLINICAL TRIAL: NCT01982916
Title: A 4 Week Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of AGR Tablet in the Treatment of Perennial Allergic Rhinitis in Korean : a Phase III Clinical Trial Bridging Study
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of AGR Tablet as a Treatment of Perennial Allergic Rhinitis in Korean
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Hospital (Other); SMG-SNU Boramae Medical Center (Other); Samsung Medical Center (Other); Kyunghee University Medical Center (Other); Konkuk University Medical Center (Other); Inha University Hospital (Other); Seoul St. Mary's Hospital (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGR_P3
Record Dates: First submitted 2013-11-07; First posted 2013-11-13 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Allergic Rhinitis; Perennial Allergic Rhinitis; Non-seasonal Allergic Rhinitis
Keywords: Allergic Rhinitis; Perennial Allergic Rhinitis; Non-seasonal Allergic Rhinitis; PAR
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AGR & Placebo (Experimental): AGR tablet by qd and Placebo by bid for 4 weeks
  Interventions: Drug: AGR tablet; Drug: Placebo (for AGR tablet and/or Active Comparator)
- Placebo (Placebo Comparator): Placebo by bid for 4 weeks
  Interventions: Drug: Placebo (for AGR tablet and/or Active Comparator)
- Active comparator (Active Comparator): Active Comparator and Placebo by bid for 4 weeks
  Interventions: Drug: Placebo (for AGR tablet and/or Active Comparator); Drug: Active Comparator

INTERVENTIONS:
Drug: AGR tablet
  Arms: AGR & Placebo
Drug: Placebo (for AGR tablet and/or Active Comparator)
Drug: Active Comparator
  Arms: Active comparator

SUMMARY:
The purpose of this study is to evaluate treatment of perennial allergic rhinitis in Korean patients with AGR tablet.

ELIGIBILITY:
Inclusion Criteria

* Males or Females no younger than 12 years.
* Patient with a history of perennial allergic rhinitis for at least an year.
* Patient with a positive prick test performed on the same day or within one year before the inclusion date.Patients had to have a (+) prick test for some allergen responsible for non-seasonal rhinitis.
* Patients with a total symptom score before the study of 5 or greater for nasal symptoms only, assessed during inclusion visit.
* Patients able to attend the required number of visits.
* A normal ECG.

Exclusion Criteria

* Patients with non-allergic rhinitis.
* Patients with obstructive nasal polyps or significant deviation of nasal septum in the investigator's criterion.
* Known hypersensitivity to tested drugs(or similar structure) or any components of the tested drugs.
* Asthmatic patients who had experienced an acute clinical attack in the three months previous to the inclusion or who had received or were receiving any type of drug for its prevention or treatment.
* Patients receiving desensitization treatment for any perennial allergen at the inclusion time. However, inclusion of subject stopping this treatment during the study period was permitted.
* Failure to pass properly the washout period of the following period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01

PRIMARY OUTCOMES:
Change of 4NTSS(4 Nasal Total Symptoms score) from baseline | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chae-Seo Rhee, M.D., Study Chair — Seoul National University Bundang Hospital; Tae-Bin Won, M.D., Principal Investigator — Seoul National University Hospital; Dae-Woo Kim, M.D., Principal Investigator — SMG-SNU Boramae Medical Center; Hyo-Yeol Kim, M.D., Principal Investigator — Samsung Medical Center; Sung-Wan Kim, M.D., Principal Investigator — Kyunghee University Medical Center; Jin-Kook Kim, M.D., Principal Investigator — Konkuk University Medical Center; Young-Hyo Kim, M.D., Principal Investigator — Inha University Hospital; Soo-Whan Kim, M.D., Principal Investigator — Seoul St. Mary's Hospital; Chang-Hoon Kim, M.D., Principal Investigator — Severance Hospital
Locations (9):
- South Korea (9):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul